CLINICAL TRIAL: NCT01888809
Title: Building Health Children: Randomized Controlled Trial (RCT) Evaluation
Brief Title: Building Healthy Children
Acronym: BHC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Monroe County Department of Human Services (Unknown); United Way of Greater Rochester (Unknown)
Responsible Party: Principal Investigator, Sheree Toth, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BHC-01
Record Dates: First submitted 2013-06-21; First posted 2013-06-28 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Teen Parenthood
Keywords: teen parents; early childhood development; home visitation; evidence-based treatment
MeSH Terms: interventions — Interpersonal Psychotherapy; Mass Screening; Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comprehensive preventive services (Experimental): Combined comprehensive services:Parents as Teachers Home visitation, Child-Parent Psychotherapy, and/or Interpersonal Psychotherapy with outreach support
  Interventions: Behavioral: Comprehensive preventive services
- Screening and referral (Active Comparator): Annual screening and referral for services as needed
  Interventions: Behavioral: Screening and referral

INTERVENTIONS:
Behavioral: Comprehensive preventive services — Combined evidence-based services:Parents as Teachers Home visitation, Child-Parent Psychotherapy, and/or Interpersonal Psychotherapy with outreach support
  Other Names: Parents as Teachers Home visitation; Child-Parent Psychotherapy; Interpersonal Psychotherapy; Outreach support
  Arms: Comprehensive preventive services
Behavioral: Screening and referral
  Arms: Screening and referral

SUMMARY:
This study will evaluate the effectiveness of providing a combination of evidence-based behavioral health treatments for mothers who gave birth to their first child prior to the age of 21 and who meet eligibility requirements and their children on prevention of child maltreatment and promotion of positive socioemotional development.

DETAILED DESCRIPTION:
Building Healthy Children is a collaboration of social service and health care agencies, each providing evidence-based services to intervention families in a seamless package. Low-income parents who gave birth to their first child when they were under 21 and who were not involved in the child welfare system were targeted as an at-risk group for whom home visitation services would offer optimal preventive and cost-efficiency outcomes. Services include Interpersonal Psychotherapy [IPT] for maternal depression and Child Parent Psychotherapy [CPP] for maternal-child relationship development and trauma treatment, and Parents As Teachers [PAT]. Families are provided a tiered complement of BHC services based upon risk and current need.

Case management and outreach services are key to assure family engagement and full program participation. An assigned community outreach worker provides a consistent, nurturing relationship that helps retain families in the program and readies parents for the evidence-based treatments, movement towards goals, and behavior change. Outreach workers help to stabilize families and ensure compliance with medical appointments and recommended care.

Most importantly, BHC home-based services are integrated with primary care practices: pediatric, family medicine, and federally qualified neighborhood health center. These comprehensive services are compared with a screening and referral only group in a randomized design. Integration with the child's medical home is an all-inclusive approach to improve child health and well-being and to achieve desired program outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include patients drawn from Strong Pediatrics, Anthony Jordan Health Center, Rochester General Hospital, or Highland Family Medicine
* residents of Monroe County,
* Temporary Assistance for Needy Families (TANF) eligible,
* are neither currently active nor have had an indicated CPS report,
* have a mother who is or was under 21 at the birth of her first child, and
* has a maximum of two children under the age of three.

Exclusion Criteria:

* Children who have indicated Child Protective reports or who are in foster care at the time of recruitment
* Any children or mothers who are not able to complete the research protocol also will be excluded.
* Potential subjects suffering from extreme medical or psychiatric conditions (such as severe brain injury or psychosis) or serious cognitive impairments (such as mental retardation) that would render them incapable of completing research measures validly will be excluded.
* Mothers with thought disorder, severe depression or suicidality requiring hospitalization, severely limited intellectual functioning (IQ less than 70), and current maternal incarceration.

Ages: 12 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1852 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Prevention of indicated Child Protective Services (CPS) reports, including change over time | Baseline and child's age of 12, 24, 36, 48, and 60 months
  Prevention of indicated Child Protective Services (CPS) reports on mothers and their children

SECONDARY OUTCOMES:
Reduction in family risks over time | Baseline and child's age of 12, 24, 36, 48, and 60 months
  Changes in family risks, including maternal depression, domestic violence exposure, health outcomes, and family stability

CONTACTS AND LOCATIONS:
Overall Officials: Sheree L Toth, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- Mt. Hope Family Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paradis HA, Sandler M, Manly JT, Valentine L. Building healthy children: evidence-based home visitation integrated with pediatric medical homes. Pediatrics. 2013 Nov;132 Suppl 2:S174-9. doi: 10.1542/peds.2013-1021R. PMID 24187121